CLINICAL TRIAL: NCT02850913
Title: Doxycycline for the Treatment of Nodding Syndrome: A Phase II, Randomised Placebo Controlled Trial
Brief Title: Doxycycline for the Treatment of Nodding Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, College of Health Sciences, Senior Lecturer, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-022; 12-16 (Other: Oxford Tropical Research Ethics Committee (OxTREC))
Record Dates: First submitted 2016-03-09; First posted 2016-08-01 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Seizures
MeSH Terms: conditions — Seizures | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxycycline (Active Comparator): * 115 participants will be randomized to oral Doxycycline 100 mg daily for six weeks.
  * Each capsule contains doxycycline hyclate equivalent to 100 mg of doxycycline base.
  * Treatment will be initiated in hospital but will be continued at home.
  * Scheduled study clinic and home visits will be conducted at 6, 12, 24 months and at 2, 4 and 6 weeks respectively for adherence monitoring and assessment of safety.
  Interventions: Drug: Doxycycline
- Placebo (Placebo Comparator): * 115 participants will be randomized to the placebo arm for matching capsules containing no active ingredients daily for six weeks.
  * Placebo will be initiated in hospital but will be continued at home.
  * Scheduled study clinic and home visits will be conducted at 6, 12, 24 months and at 2, 4 and 6 weeks respectively for adherence monitoring and assessment of safety.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Doxycycline — * 115 participants will be randomized to either oral Doxycycline 100 mg daily for six weeks.
  * Treatment will be initiated in hospital but will be continued at home.
  * Scheduled study clinic visits will be made by the participants at 6, 12 and 24 months.
  * Each participant will be visited at home at 2, 4 and 6 weeks for adherence monitoring and assessment of safety
  Other Names: Doxycycline hyclate
  Arms: Doxycycline
Other: Placebo — - Placebo (matching capsules containing no active ingredients)
  Arms: Placebo

SUMMARY:
Nodding syndrome (NS) is a devastating neurologic disorder affecting thousands of children in Africa. A number of toxic, nutritional, infectious, para-infectious and environmental causes have been studied but the only consistent association has been with infection by the parasite Onchocerca volvulus. There is no specific treatment for NS and also for the adult onchocerca. However, antibiotic depletion of the Onchocerca volvulus co-symbiotic bacteria Wolbachia with tetracyclines such as doxycycline results in sterilisation and premature death of the adult worm and marked reductions in dermal microfilaria density. Potentially, such therapy that kills adult onchocerca volvulus may improve the outcome of NS if the association were true.

DETAILED DESCRIPTION:
Primary hypothesis

Oral doxycycline 100mg daily for six weeks in patients with NS aged 8 years or older will reduce inflammatory responses and the proportion of patients with serum antibodies to NSPs or leiomodin 24 months after intervention by 40% compared to placebo.

Primary efficacy objective

To determine the effects of doxycycline 100mg daily for six weeks in patients with NS 8 years or older on serum levels of antibodies to NSPs (VGKC complex and others to be identified in a concurrent case-control study) or leiomodin at 24 months.

Study Type

This will be a two-arm, placebo-controlled (double blind) randomized phase II trial of oral doxycycline 100mg daily for six weeks.

Study site

Kitgum general hospital, Kitgum, Uganda.

Study Population

Study participants will be patients with confirmed NS as defined according to the World Health Organization (WHO) consensus case definition i.e. (i) Head nodding on two or more occasions, (ii) Occurring in clusters at a frequency of 5-20/minute, (iii) Onset between the ages of 3-18 years, (iv) Observed by a trained health worker or documented on EEG

Plus any one of:

a) triggered by food or cold weather; b) presence of other seizures or neurological abnormalities and cognitive decline and c) clustering in space or time), age ≥8 years, and with written consent from a parent or guardian.

Study Interventions

Participants will receive standard of care supportive treatment according to current guidelines for NS (antiepileptic drug treatment with sodium valproate, management of psychiatric disorders, nutritional, physical and occupational therapy as indicated).

All will be hospitalised in the first weeks during which period, baseline measurements including clinical assessments, EEG, cognitive and laboratory testing will be performed and antiepileptic drug doses rationalised.

Sample size: The sample size (115 participants per arm i.e. 230 total) is estimated based on the assumption that a six-weeks treatment course of doxycycline will reduce the proportion of participants with antibodies to NSPs or Leiomodin by 40% (from 50.0% to 30.0%) 24 months after initiation of the intervention while providing for 10% loss to follow-up (β=80%, α=0.05).

Participants will then be randomised to either oral doxycycline (Azudox®, Kampala Pharmaceutical Industries, Ltd) 100mg daily for six weeks or identical placebo. Treatment will be initiated in hospital but will be continued at home. Each participant will be visited at home at 2, 4 and 6 weeks for adherence monitoring and assessment of safety and will report back to the hospital study clinic at 6, 12 and 24 months.

Follow-up procedures:

Participants will be followed up at 2, 4, and 6 weeks by the health visitor to document adherence and assess safety and will be assessed for outcomes in hospital at 24 months after initiation of the intervention.

Data Analysis:

Primary analysis will be by intention to treat. The investigators will examine the effect of doxycycline at 24 months on antibodies to host NSPs and leiomodin, inflammatory responses (CRP, C3a and C3b), on epileptiform discharges and seizure control, and microfilaria density/ Wolbachia load, and on clinical (cognitive, motor, psychiatric and quality of life) symptoms compared to placebo.

In a sub-analysis, the investigators will examine the effects of the intervention in new patients compared to patients with long standing symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with confirmed NS as defined by the WHO i.e. Head nodding on two or more occasions (both past and current)

   * Symptom onset between the ages of 3-18 years
   * Observed by a trained health worker or documented on EEG

   Plus any one of:
   * Triggered by food or cold weather
   * Presence of other seizures or neurological abnormalities and cognitive decline
   * Clustering in space or time.
2. Age 8 years or older
3. Written consent by the parent or guardian

Exclusion Criteria:

1. Females with a positive urinary HCG (pregnancy) test
2. Patients receiving Phenobarbitone, Carbamazepine, Phenytoin or Rifampicin.
3. Known hypersensitivity to study drug
4. Withdrawal of consent since enrollment
5. Reported inability to swallow capsules
6. Enrolled or known agreement to enroll into another clinical trial involving ongoing or scheduled treatment with medicinal products during the course of the study
7. Suspected high likelihood of non-compliance with study drug and the follow-up schedule - e.g. dependent on a carer who is unlikely to consistently be available.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 230 (Estimated)
Dates: Start 2016-09-05 (Actual); Primary Completion 2020-04-05 (Estimated); Study Completion 2020-08-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with antibodies to Neuron Surface Proteins (NSPs) or leiomodin at 24 months. | 24 months

SECONDARY OUTCOMES:
Mean change in serum concentrations of antibodies to NSPs or leiomodin | From baseline (time 0 months) to 24 months
Mean change in serum concentrations of C-Reactive Protein | From baseline (time 0 months) to 24 months
Mean change in serum concentrations of C3a and C3b | From baseline (time 0 months) to 24 months
Mean change in dermal microfilaria density on real time Polymerase Chain Reaction at 24 months | From baseline (time 0 months) to 24 months
The proportions of patients achieving seizure freedom (≥1 month without head nodding or convulsive seizures) | 24 months
Proportion of patients with interictal epileptiform discharges on 30-minute diagnostic EEG | 24 months
Proportion of participants with Gross Motor Function Classification System (GMFCS) scores 3-5 | 24 months
Proportion of participants with mental health disorders on the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) | 24 months
Mean change in cogstate scores | From baseline (time 0 months) to 24 months
Proportion of participants with improved Quality of Life (a perception) on the Quality of Life in Childhood Epilepsy Questionnaire | From baseline (time 0 months) to 24 months
Incidence rate of non-nodding syndrome sick clinic visits and all cause sick clinic visits | 24 months
The proportion of participants with stunting (height for age Z-scores <-3 SD) | 24 months
The proportion of participants with wasting (weight for height Z-scores <-3 SD) | 24 months
All-cause mortality | 24 months
Incidence rate of all-cause hospital admissions | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Idro, MMED, PhD, Principal Investigator — Makerere University College of Health Sciences; Kevin Marsh, MRCP, DTM&H, Principal Investigator — University of Oxford
Locations (1):
- Makerere University College of Health Sciences, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Idro R, Ogwang R, Anguzu R, Akun P, Ningwa A, Abbo C, Giannoccaro MP, Kubofcik J, Mwaka AD, Nakamya P, Opar B, Taylor M, Nutman TB, Elliott A, Vincent A, Newton CR, Marsh K. Doxycycline for the treatment of nodding syndrome: a randomised, placebo-controlled, phase 2 trial. Lancet Glob Health. 2024 Jul;12(7):e1149-e1158. doi: 10.1016/S2214-109X(24)00102-5. Epub 2024 May 13. PMID 38754459
- [Derived] Idro R, Anguzu R, Ogwang R, Akun P, Abbo C, Mwaka AD, Opar B, Nakamya P, Taylor M, Elliott A, Vincent A, Newton C, Marsh K. Doxycycline for the treatment of nodding syndrome (DONS); the study protocol of a phase II randomised controlled trial. BMC Neurol. 2019 Mar 6;19(1):35. doi: 10.1186/s12883-019-1256-z. PMID 30841858
- [Derived] Anguzu R, Akun PR, Ogwang R, Shour AR, Sekibira R, Ningwa A, Nakamya P, Abbo C, Mwaka AD, Opar B, Idro R. Setting up a clinical trial for a novel disease: a case study of the Doxycycline for the Treatment of Nodding Syndrome Trial - challenges, enablers and lessons learned. Glob Health Action. 2018;11(1):1431362. doi: 10.1080/16549716.2018.1431362. PMID 29382251